CLINICAL TRIAL: NCT03831971
Title: The Influence of ANS-6637 on Midazolam Pharmacokinetics in Healthy Volunteers (SEARCH PK)
Brief Title: The Influence of ANS-6637 on Midazolam Pharmacokinetics in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 190052; 19-CC-0052
Record Dates: First submitted 2019-02-05; First posted 2019-02-06 (Actual); Results first posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2019-12-30

CONDITIONS: Opiod Use Disorder
Keywords: Reward Pathway; Pharmacokinetics; Dopamine; Opioid Use; Addiction
MeSH Terms: conditions — Behavior, Addictive | interventions — ANS-6637

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ANS-6637 & Midazolam (Experimental): Subjects will receive (1) midazolam 5 mg po single dose on Day 1 followed by (2) Drug free period on Day 2 followed by (3) ANS-6637 600 mg po daily (Days 3-7) to reach steady state followed by (4) ANS-6637 600 mg po single dose + midazolam 5mg po single dose on Day 8
  Interventions: Drug: ANS-6637

INTERVENTIONS:
Drug: ANS-6637 — Subjects will receive (1) midazolam 5 mg po single dose on Day 1 followed by (2) Drug free period on Day 2 followed by (3) ANS-6637 600 mg po daily (Days 3-7) to reach steady state followed by (4) ANS-6637 600 mg po single dose + midazolam 5mg po single dose on Day 8

SUMMARY:
Background:

Opioids are medicines that control pain. But they are often misused, which can lead to illness and death. Opioids increase dopamine to the brain, which makes people feel good and often causes them to crave drugs, leading to misuse and addiction. An investigational drug ANS-6637 may lower the dopamine surge and stop opioid craving. Midazolam is a drug approved for anxiety. Researchers want to give the two drugs together and see if ANS-6637 affects midazolam levels, to help understand how ANS-6637 is used in the body.

Objective:

To study the safety, tolerability, and effects of ANS-6637 taken with and without midazolam.

Eligibility:

Healthy adults 18 65 years old

Design:

Participants will be screened with a medical history, physical exam, and blood and heart tests. Participants who can get pregnant will have a pregnancy test.

Participants must agree to use 2 types of birth control during the study, if applicable.

Participants will stay at the clinic for 10 days. Meals will be provided. Participants will not be allowed to:

Leave NIH campus

Eat or drink anything with caffeine, alcohol, or certain juices

Use any nicotine or related products (including vaping)

Use any medicines (including herbal)

During the clinic stay, participants will:

Fast overnight several times

Have blood drawn most days. Twice, a small tube will be inserted in an arm vein for frequent blood samples.

Repeat screening tests and answer questions about their mood several times

Get midazolam syrup in water on 1 day

Take 6 ANS-6637 tablets by mouth on 5 days

Take both study drugs on 1 day

A few days later, participants will have a follow-up visit to repeat screening tests and answer questions about their mood.

DETAILED DESCRIPTION:
Opioid use causes a myriad of effects which contribute to significant morbidity and early mortality, and is associated with risky sexual behavior and injection drug use (IDU), two major forms of human immunodeficiency virus (HIV) and hepatitis C virus (HCV) transmission in urban and suburban United States. Through these high-risk behaviors, persons with opioid use disorder (OUD) develop both direct comorbidities (e.g. blood stream infections and infectious endocarditis), as well as risk-associated illnesses (e.g. sexually transmitted infections, HCV and hepatitis B virus [HBV]) which have considerable downstream health care effects. As such, there is a need for pharmacologic agents in the treatment of OUD that go beyond avoidance of withdrawal and facilitate decreased frequency or complete cessation of opioid use.

The biologic mechanism of OUD, common to all forms of addiction, is a conditioned drug cue-related response in the CNS, causing a dopamine surge. If effective, a central pharmacologic strategy targeting the aberrant reward circuitry seen in OUD could potentially reduce drug craving and result in opioid abstinence.

In the SEARCH Pharmacokinetic (PK) investigation, we aim to understand the pharmacokinetic signal of the novel, oral agent ANS-6637, an aldehyde dehydrogenase 2 (ALDH-2) inhibitor that has the potential to reduce dopamine surge in the CNS and inhibit opioid craving. In preclinical studies, the active metabolite of ANS-6637, GS-548351, showed substrate dependent inhibition of CYP3A in vitro, with little or no inhibitory effect on the activities of other cytochrome P450 (CYP) enzymes. As such, the current investigation seeks to explore the potential inhibition of CYP3A by ANS-6637 with the FDA-recommended CYP3A probe substrate, midazolam.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Must have the ability to understand and must personally sign a written informed consent form, which must be obtained prior to initiation of study procedures.
2. Must be between 18 and 65 years of age, inclusive.
3. Must have discontinued use of nicotine and nicotine containing products including vaping or juuling from 90 days prior to study drug dosing and throughout the study duration.
4. Must be willing to abstain from any food or beverages containing alcohol 72 hours prior to first dose and through follow-up visit.
5. Must be willing to abstain from cannabis 72 hours prior to first dose and through follow-up visit.
6. Must be willing to abstain from caffeine (including tea, coffee, chocolate) or grapefruit, Seville orange juice or other methyl xanthine containing foods (e.g. theophylline, theobromine, tea leaves, yerba mate, kola nuts and guarana berries) 72 hours prior to the first dose and through follow- up visit.
7. Must have a body mass index (BMI) from 19 to 30 kg/m^2 (inclusive) at screening.
8. Must be human immunodeficiency virus type 1 (HIV-1) antibody negative at screening.
9. Must be hepatitis B (HBV) surface antigen negative at screening.
10. Must be hepatitis C (HCV) antibody or RNA negative at screening.
11. Male subjects must refrain from sperm donation from clinic admission, throughout the study period, and continuing for at least 90 days following the last dose of study drug.
12. Subjects must refrain from blood donation from clinic admission, throughout the study period, and continuing for at least 30 days following the last dose of study drug.
13. Must be willing to comply with contraception guidelines below Contraception:

    The fetal risks associated with ANS-6637 are not known, but pre- clinical animal data demonstrate some risk. Subjects must agree not to become pregnant or impregnate a female. Females of childbearing potential must have a reproductive risk assessment done to determine the risk of undetectable pregnancy at study start [i.e. sexual and contraceptive history for 30 days preceding screening] pregnancy test at screening and baseline (Day 0). For the duration of the study, subject and their partners must practice two non-hormonal methods of birth control, having begun no less than 30 days, without interruption, prior to screening. They must continue to use both methods until 3 months after stopping the study drug. Two of the three methods of birth control listed below MUST be used, or an alternative combination offering very high efficacy, per the PI, in consultation with the Sponsor Medical Monitor may be considered:
    * Male or female condoms [but not both] with a spermicide
    * Diaphragm with a spermicide
    * Intrauterine device (IUD)

    If pregnancy is suspected or should occur, subjects must notify the study staff immediately.
14. Must, in the opinion of the Investigator, be in good health based upon medical history and physical examination, and screening laboratory evaluations.
15. Judged to be healthy based on medical history, physical examination, vital signs, and clinical laboratory tests at screening and Day 0: liver function tests (AST, ALT, Tbili) less than or equal to upper limit of normal [ULN], platelets (PLT) >150,000/ microliter, hemoglobin (Hgb) >13 g/dL (males); >12 g/dL (females), CK less than or equal to 2x ULN, Amylase/lipase < ULN, thyroid function tests [TSH and T4] within normal range, fasting total cholesterol <240 mg/dL, or fasting triglycerides <240 mg/dL, per DAIDS AE table and Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Trials AE table for total bilirubin [Tbili] only.
16. Must be willing and able to comply with all study requirements.

EXCLUSION CRITERIA:

1. Therapy with any prescription, over-the-counter (OTC), herbal, or holistic medications, including hormonal contraceptives by any route, within 5 half- lives of the agent prior to receipt of any study medications will not be permitted with the following exception: Intermittent or short-course therapy (<14 days) with prescription or OTC medications, herbals, or holistic medications within the screening period prior to starting study drugs may be permitted after review by the investigators on a case-by-case basis for potential drug interactions. Receipt of influenza vaccination will be allowed prior to, during, and/or after the study.
2. Have any serious or active medical, surgical, or psychiatric conditions which, in the opinion of the Investigator, would interfere with subject treatment, assessment, or compliance with the protocol.
3. Have previously participated in an investigational trial involving administration of any investigational compound within 30 days prior to screening.
4. Have current, or a history of mild to severe alcohol use, cannabis or other substance use disorder including any use of illicit drugs as defined by DSM-5 criteria, within 12 months of first study dose
5. Renal impairment (chronic renal insufficiency of any chronic kidney disease stage, or acute renal failure not induced by drug therapy defined as eGFR <90 ml/min)
6. Have a positive urine drug test (ethanol, cannabis, barbiturates, cocaine, opiates, or amphetamines) at Screening or Day 0.
7. History of flushing or intolerance related to alcohol consumption using the NIAAA screening assessment questionnaire tool for alcohol flushing
8. Inability to obtain venous access for sample collection.
9. Have a history of significant drug sensitivity or drug allergy to any benzodiazepines.
10. Known hypersensitivity to formulation excipients: microcrystalline cellulose, croscarmellose sodium, magnesium stearate, polyvinyl alcohol, titanium dioxide, polyethylene glycol, and talc.
11. Have been treated with systemic steroids, immunosuppressant therapies or chemotherapeutic agents within 3 months of study screening or expected to receive these agents during the study (e.g., corticosteroids, immunoglobulins, and other immune- or cytokine-based therapies).
12. Presence or history of clinically significant cardiovascular disease, cardiomyopathy, and/or cardiac conduction abnormalities.
13. Have clinically significant ECG abnormalities or any of the following ECG abnormalities at Screening: PR >220 msec; QRS >120 msec; QTcF >450 msec; HR <40 beats per minute; second or third degree heart block.
14. Have a history or family history of Long QT Syndrome, Brugada syndrome, Wolfe-Parkinson-White Syndrome, or have a family history of sudden cardiac death or unexplained death in an otherwise healthy individual between the ages of 1 and 30 years.
15. Have history of syncope, palpitations, unexplained dizziness or chronic nausea or headaches.
16. Have an implanted defibrillator or pacemaker.
17. Have a history of liver disease, including Gilbert's Disease.
18. Any clinically significant electrolyte abnormality (outside of NIH normal reference ranges) at screening (e.g., hypokalemia, hypocalcemia, hypomagnesemia) or any condition that could lead to abnormal electrolyte disturbances (eg, eating disorder).
19. Have a history of taking dopamine antagonists/anti-psychotics.
20. Are unable to comply with study requirements.
21. Positive urine toxicology screen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Masur, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diamond I, Yao L. From Ancient Chinese Medicine to a Novel Approach to Treat Cocaine Addiction. CNS Neurol Disord Drug Targets. 2015;14(6):716-26. doi: 10.2174/1871527314666150529144329. PMID 26022266
- [Background] Yao L, Fan P, Arolfo M, Jiang Z, Olive MF, Zablocki J, Sun HL, Chu N, Lee J, Kim HY, Leung K, Shryock J, Blackburn B, Diamond I. Inhibition of aldehyde dehydrogenase-2 suppresses cocaine seeking by generating THP, a cocaine use-dependent inhibitor of dopamine synthesis. Nat Med. 2010 Sep;16(9):1024-8. doi: 10.1038/nm.2200. Epub 2010 Aug 22. PMID 20729865
- [Background] Volkow ND, Koob GF, McLellan AT. Neurobiologic Advances from the Brain Disease Model of Addiction. N Engl J Med. 2016 Jan 28;374(4):363-71. doi: 10.1056/NEJMra1511480. No abstract available. PMID 26816013
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-CC-0052.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 26 subjects signed consent. 14 subjects not eligible. 12 subjects underwent study.
Period: Overall Study
Arm/Group | ANS-6637 & Midazolam
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ANS-6637 & Midazolam
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 6
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics - Time to Maximum Concentration of Midazolam Alone
Description: Time to maximum plasma concentration (tmax). The summary PK results were informed by a continuous measurement at the following serial blood collection time points: 0 (pre-dose), then 0.5, 1, 2, 3, 4, 6, 8, 12, 22, and 24 hours postdose.
Time Frame: Day 1
Population: Participants who received midazolam
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | ANS-6637 & Midazolam
Number analyzed (Participants) | 12
hours | 0.58 (55.4)

2. Primary Outcome: Pharmacokinetics - Time to Maximum Concentration of 1-hydroxymidazolam Alone
Description: as for outcome 1
Time Frame: Day 1
Population: Participants who received midazolam
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | ANS-6637 & Midazolam
Number analyzed (Participants) | 12
hours | 0.58 (55.4)

3. Primary Outcome: Pharmacokinetics - Maximum Total Plasma Concentration of Midazolam Alone
Description: Maximum total plasma concentration (Cmax). The summary PK results were informed by a continuous measurement at the following serial blood collection time points: 0 (pre-dose), then 0.5, 1, 2, 3, 4, 6, 8, 12, 22, and 24 hours postdose.
Time Frame: Day 1
Population: Participants who received midazolam
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ANS-6637 & Midazolam
Number analyzed (Participants) | 12
ng/mL | 14.28 (46.5)

4. Primary Outcome: Pharmacokinetics - Maximum Total Plasma Concentration of 1-hydroxymidazolam Alone
Description: as for outcome 3
Time Frame: Day 1
Population: Participants who received midazolam
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ANS-6637 & Midazolam
Number analyzed (Participants) | 12
ng/mL | 9.04 (65.3)

5. Primary Outcome: Pharmacokinetics - Plasma Exposure of Midazolam Alone
Description: Midazolam plasma area under the concentration time curve 0-infinity. The summary PK results were informed by a continuous measurement at the following serial blood collection time points: 0 (pre-dose), then 0.5, 1, 2, 3, 4, 6, 8, 12, 22, and 24 hours postdose.
Time Frame: Day 1
Population: Participants who received midazolam
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng * h/mL
Arm/Group | ANS-6637 & Midazolam
Number analyzed (Participants) | 12
ng * h/mL | 49.73 (58.8)

6. Primary Outcome: Pharmacokinetics - Plasma Exposure of 1-hydroxymidazolam Alone
Description: 1-hydroxymidazolam plasma area under the concentration time curve (time 0-infinity). The summary PK results were informed by a continuous measurement at the following serial blood collection time points: 0 (pre-dose), then 0.5, 1, 2, 3, 4, 6, 8, 12, 22, and 24 hours postdose.
Time Frame: Day 1
Population: Participants who received midazolam
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng * h/mL
Arm/Group | ANS-6637 & Midazolam
Number analyzed (Participants) | 12
ng * h/mL | 27.2 (59.3)

7. Primary Outcome: Pharmacokinetics - Elimination of Midazolam Alone
Description: Half-life. The summary PK results were informed by a continuous measurement at the following serial blood collection time points: 0 (pre-dose), then 0.5, 1, 2, 3, 4, 6, 8, 12, 22, and 24 hours postdose.
Time Frame: Day 1
Population: Participants who received midazolam
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | ANS-6637 & Midazolam
Number analyzed (Participants) | 12
hours | 4.68 (23.3)

8. Primary Outcome: Pharmacokinetics - Elimination of 1-hydroxymidazolam Alone
Description: as for outcome 7
Time Frame: Day 1
Population: Participants who received midazolam
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | ANS-6637 & Midazolam
Number analyzed (Participants) | 12
hours | 5.29 (31.8)

9. Primary Outcome: Pharmacokinetics - Time to Maximum Concentration of Midazolam: Midazolam Plus Steady State ANS-6637
Description: as for outcome 1
Time Frame: Day 8
Population: Participants who received midazolam and ANS-6637
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | ANS-6637 & Midazolam
Number analyzed (Participants) | 12
hours | 0.69 (87.8)

10. Primary Outcome: Pharmacokinetics - Time to Maximum Concentration of 1-hydroxymidazolam: Midazolam Plus Steady State ANS-6637
Description: as for outcome 1
Time Frame: Day 8
Population: Participants who received midazolam and ANS-6637
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | ANS-6637 & Midazolam
Number analyzed (Participants) | 12
hours | 0.69 (87.8)

11. Primary Outcome: Pharmacokinetics - Maximum Total Plasma Concentration of Midazolam: Midazolam Plus Steady State ANS-6637
Description: as for outcome 3
Time Frame: Day 8
Population: Participants who received midazolam and ANS-6637
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ANS-6637 & Midazolam
Number analyzed (Participants) | 12
ng/mL | 17.47 (37)

12. Primary Outcome: Pharmacokinetics - Maximum Total Plasma Concentration of 1-hydroxymidazolam: Midazolam Plus Steady State ANS-6637
Description: as for outcome 3
Time Frame: Day 8
Population: Participants who received midazolam and ANS-6637
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ANS-6637 & Midazolam
Number analyzed (Participants) | 12
ng/mL | 8.61 (59.3)

13. Primary Outcome: Pharmacokinetics - Plasma Exposure of Midazolam: Midazolam Plus Steady State ANS-6637
Description: as for outcome 5
Time Frame: Day 8
Population: Participants who received midazolam and ANS-6637
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng * h/mL
Arm/Group | ANS-6637 & Midazolam
Number analyzed (Participants) | 12
ng * h/mL | 62.63 (46.7)

14. Primary Outcome: Pharmacokinetics - Plasma Exposure of 1-hydroxymidazolam: Midazolam Plus Steady State ANS-6637
Description: 1-hydroxymidazolam plasma area under the concentration time curve 0-infinity. The summary PK results were informed by a continuous measurement at the following serial blood collection time points: 0 (pre-dose), then 0.5, 1, 2, 3, 4, 6, 8, 12, 22, and 24 hours postdose.
Time Frame: Day 8
Population: Participants who received midazolam and ANS-6637
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng * h/mL
Arm/Group | ANS-6637 & Midazolam
Number analyzed (Participants) | 12
ng * h/mL | 29.28 (53.3)

15. Primary Outcome: Pharmacokinetics - Elimination of Midazolam: Midazolam Plus Steady State ANS-6637
Description: as for outcome 7
Time Frame: Day 8
Population: Participants who received midazolam and ANS-6637
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | ANS-6637 & Midazolam
Number analyzed (Participants) | 12
hours | 4.64 (20.1)

16. Primary Outcome: Pharmacokinetics - Elimination of 1-hydroxymidazolam: Midazolam Plus Steady State ANS-6637
Description: as for outcome 7
Time Frame: Day 8
Population: Participants who received midazolam and ANS-6637
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | ANS-6637 & Midazolam
Number analyzed (Participants) | 12
hours | 5.76 (34.6)

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | ANS-6637 & Midazolam
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ANS-6637 & Midazolam (N=12)
Dizziness (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 3
Fatigue (General disorders) | 12
Pain (General disorders) | 1
Bacteriuria (Infections and infestations) | 3
Alanine aminotransferase increased (Investigations) | 1
Amylase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood bicarbonate abnormal (Investigations) | 1
Blood cholesterol increased (Investigations) | 4
Blood creatinine increased (Investigations) | 1
Creatinine renal clearance decreased (Investigations) | 5
Electrocardiogram PR prolongation (Investigations) | 1
Urine analysis abnormal (Investigations) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Insomnia (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT03831971/Prot_SAP_000.pdf